CLINICAL TRIAL: NCT06038344
Title: Evaluation of the Gluten Free Food Guide on Diet Quality and Adherence to the GFD in Newly Diagnosed Children and Youth With Celiac Disease in the Clinical Setting
Brief Title: Influence of a Gluten Free Food Guide on Diet Quality and Adherence to the GFD in Youth With Celiac Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00111071
Record Dates: First submitted 2023-08-29; First posted 2023-09-14 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Celiac Disease in Children; Gluten Enteropathy; Diet; Deficiency; Adherence, Treatment
Keywords: Gluten-Free Food Guide; Dietary Education; Dietary Quality; Celiac Disease
MeSH Terms: conditions — Celiac Disease; Malnutrition; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care + Gluten-free food guide teaching (Experimental): 45-minute dietary counselling session using the novel gluten-free food guide conducted by a researcher over Zoom. This occurs after standard of care dietary education by an RD. The gluten free teaching session in the study protocol focuses on the GF plate model, the rationale for the GF plate model, and addressing the individual participants dietary needs based on a dietary intake assessment by a trained investigator using specific educational materials that are present in the guide.
  Interventions: Behavioral: Gluten-free food guide teaching
- Standard of Care (No Intervention): 45-minute group session on the gluten-free diet conducted by registered dietitians over Zoom. The registered dietitian's dietary education included a virtual group class focusing on gluten literacy, meal planning, food label reading and dietary intake based on Canada's Food Guide to Healthy Eating (2019).

INTERVENTIONS:
Behavioral: Gluten-free food guide teaching — Teaching the gluten-free food guide will be done over Zoom within 1-2 weeks of the dietitian's standard of care teaching (group Zoom session). This teaching will take 30-45 minutes and will be conducted by a trained researcher. The investigators will use the gluten-free food guide as teaching materials with a focus on the GF plate model, the rationale for the GF plate model, nutritional consideration of gluten-free diet and content related to the additional 24 teaching materials (e.g. folate, fibre, eating out, school lunches etc.) contained within the guide. Individualized dietary suggestions based on participants' food records will also be provided.
  Arms: Standard of Care + Gluten-free food guide teaching

SUMMARY:
Celiac disease (CD) is an autoimmune gastrointestinal disease that is caused by intolerance to gluten in the diet. The mainstay of treatment is a gluten-free diet (GFD). Children with CD on the GFD often have low micronutrient intakes (e.g. folate, iron) and high intakes of sugar and fat. Current Canadian nutrition guideline does not address these nutritional limitations. The investigation team developed a novel GF-food guide (GFFG). This randomized clinical trial aims to evaluate the impact of GFFG on diet quality and adherence to the GFD in newly diagnosed children and youth with celiac disease in the clinical setting. The investigators will compare dietary counselling using the GFFG versus the standard of care in children newly diagnosed with CD and their parents to see if participant care outcomes (diet quality, nutrition literacy, adherence to the GFD) improved over six months.

DETAILED DESCRIPTION:
Background: The only treatment for celiac disease (CD) is the gluten-free (GF) diet which affects every 1 in 100 individuals. Non-adherence to the diet can lead to intestinal damage and nutrient malabsorption, which can negatively impact a critical period of growth and development in children. Despite adherence, the GF diet does not guarantee nutritional adequacy in children and can lead to obesity and chronic disease. A number of studies confirm that children and adults on GFDs often face several nutritional challenges, including low intakes of fibre, vitamin D, zinc, magnesium and high intakes of simple sugars and saturated fats associated with poor diet quality. Prepackaged GF foods are often high in simple sugars and saturated fat while being low in fibre, which are all known risk factors for the development of chronic disease in the adult population. While parents and newly diagnosed children with CD show significant improvements in knowledge about the GF diet after receiving standard-of-care education from healthcare practitioners at the time of diagnosis, some children with CD continue to experience significant challenges with reduced diet quality and nutritional inadequacy while on the GF diet, even after dietary education. Currently, there are no existing nutrition guidelines that are focused on the GFD. To address this issue, the investigation team recently developed a gluten-free food guide (GFFG). The GFFG consists of overall diet recommendations with a layout that mirrors the new Canada's Food Guide, associated teaching materials that address concepts related to nutrition literacy and knowledge as identified in the pre-guide stakeholder engagement with health care providers (RD, RN, MD) and families with children with CD (Mager et al., Br J Nutr 2022). Focus groups and online surveys were conducted for feasibility analysis with end-stakeholders (health professionals, parents/caregivers of children with CD, and adolescents with CD) to enable a comprehensive evaluation of the feasibility of the food guide in terms of content and layout (Mager et al., Br J Nutr 2022).

Study Objective: The study purpose is to compare the impact of dietary counselling using the GFFG versus standard of care (SOC) in children/adolescents and their parent/caregiver newly diagnosed with CD on participant care outcomes (diet quality, nutrition literacy, adherence to the GFD) over six months.

Hypothesis: The GFFG will increase diet quality and parental food literacy and improve adherence to the GFD in newly diagnosed children with CD and their parents over six months.

Sample size: Forty families (20/group) are proposed to enroll in this study. This sample size was based on a convenient sample.

Data Analysis: Data will be expressed as mean (± SD) or median (interquartile range) for parametric and non-parametric variables, respectively (tested by the Shapiro-Wilk test). T-tests (parametric) or Mann Whitney (non-parametric) tests to compare household characteristics (sociodemographic), adherence to the GFD, and DQ between SOC vs SOC+GFFG. Pearson and/or Spearman correlations will be conducted to assess the associations between child DQ and parental nutrition literacy, GFD adherence and household sociodemographics. Chi-square tests will be used to determine significant differences between categorical variables. P value < 0.05 adjusted for multiple comparisons will determine statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents, male and female, 5-18 years of age and their parents.
* Clinically diagnosed celiac disease
* Diagnosis within 3 months

Exclusion Criteria:

* Children, male and female, <5 years of age
* Celiac disease diagnosis >3 months
* Children/adolescents diagnosed with type 1 diabetes (T1D)
* Not clinically diagnosed with celiac disease

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Dietary quality | Baseline
  Child/adolescent dietary intake will be collected using three-day food intake records (2 weekdays and 1 weekend day), and diet quality will be analyzed using Healthy Eating Index-Canada (score out of 100) at study entry. The maximum score for Healthy Eating Index-Canada is 100 (indicating high diet quality) and the lowest score of 0 reflects poor diet quality. Scores of 80 and over are representative of good-excellent diet quality, Scores of 60-80 reflect needs improvement of diet quality and less than 60 indicative of poor diet quality.
Dietary quality | 6 months
  Child/adolescent dietary intake will be collected using three-day food intake records (2 weekdays and 1 weekend day), and diet quality will be analyzed using Healthy Eating Index-Canada (score out of 100) at 6 months. The maximum score for Healthy Eating Index-Canada is 100 (indicating high diet quality) and the lowest score of 0 reflects poor diet quality. Scores of 80 and over are representative of good-excellent diet quality, Scores of 60-80 reflect needs improvement of diet quality and less than 60 indicative of poor diet quality.

SECONDARY OUTCOMES:
Self-reported adherence to the gluten-free diet. | Baseline
  Assessment of child/adolescent adherence to the GFD will be evaluated by a self-reported questionnaire (Kindl Test ®) at baseline. This is a questionnaire that consists of 10 questions related to dietary adherence and quality of life. Max score is 10. Minimum score is 0. Higher scores indicative of lower adherence and quality of life.
Self-reported adherence to the gluten-free diet | 6 months
  Assessment of child/adolescent adherence to the GFD will be evaluated by a self-reported questionnaire (Kindl Test ®) at 6 months. This is a questionnaire that consists of 10 questions related to dietary adherence and quality of life. Max score is 10. Minimum score is 0. Higher scores indicative of lower adherence and quality of life.
Gluten intake | Baseline
  Assessment of changes in child/adolescent gluten intake will be calculated from a 3-day food record using the gluten-calculation equation ((grain weight (in gms) *20)/1000) at study entry. Gluten Values less than 10 mg/d in the diet considered low gluten intake associated with adherence to the gluten free diet.
Gluten intake | 6 months
  Assessment of changes in child/adolescent gluten intake will be calculated from a 3-day food record using the gluten-calculation equation ((grain weight (in gms) *20)/1000)at 6 months. Gluten Values less than 10 mg/d in the diet considered low gluten intake associated with adherence to the gluten free diet.
Parental Nutrition Literacy | Baseline
  Parental nutrition literacy will be measured using the validated Nutrition Literacy Assessment Tool for Adults at study entry. The validated tool consists of 30 questions and scoring can range between 0-30. Excellent scores > 24.
Parental Nutrition Literacy | 6 months
  Parental nutrition literacy will be measured using the validated Nutrition Literacy Assessment Tool for Adults at six months. The validated tool consists of 30 questions and scoring can range between 0-30. Excellent scores > 24.

CONTACTS AND LOCATIONS:
Overall Officials: Diana R Mager, Principal Investigator — University of Alberta
Locations (1):
- Clinical Research Unit, University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Data will only be presented in aggregate form in peer review publications and/or conference proceedings.

REFERENCES:
- [Background] Mager DR, Cyrkot S, Lirette C, Brill H, Dowhaniuk J, Mileski H, Basualdo-Hammond C, Nasser R, Assor E, Marcon M, Turner JM. Nutritional considerations of a paediatric gluten-free food guide for coeliac disease. Br J Nutr. 2022 Feb 14;127(3):421-430. doi: 10.1017/S0007114521000994. Epub 2021 Mar 22. PMID 33745459
- [Background] Mager DR, Cyrkot S, Lirette C, Brill H, Dowhaniuk J, Mileski H, Basualdo-Hammond C, Nasser R, Assor E, Marcon M, Turner JM. Evaluation of a paediatric gluten-free food guide by children and youth with coeliac disease, their parents and health care professionals. Br J Nutr. 2022 Jun 28;127(12):1784-1795. doi: 10.1017/S0007114521002774. Epub 2021 Jul 23. PMID 34294170